CLINICAL TRIAL: NCT02243852
Title: Evaluation of the Effects of Growth Hormone (GH) Deficiency and Growth Hormone Replacement on Serum Fibroblast Growth Factor 21 (FGF21) Concentration in Patients with Growth Hormone Deficiency (GHD)
Brief Title: Effects of Growth Hormone (GH) Deficiency and Growth Hormone Replacement on Serum Fibroblast Growth Factor 21 (FGF21)
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor withdrew support 6th June 2017
Sponsor: University of Liverpool (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 13/NW/0075
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2014-09

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Hormone Deficiency (GHD); Growth Hormone Replacement Therapy; Fibroblast Growth Factor 21 (FGF21); Visceral Fat; Subcutaneous Fat
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All patients will have a 15 ml blood sample taken for glucose, insulin, lipid profile and liver function tests (LFTs). Insulin sensitivity will be measured by HOMA-IR. Plasma concentrations of FGF-21 will be measured using a commercial ELISA kit (Human FGF-21; Biovendor, Germany).
  16 GHD patients, who are eligible for GH replacement therapy as part of their routine clinical care, according to the National Institute for Clinical Excellence (NICE) recommendations, based on the biochemical deficiency and the appropriate AGHDA questionnaire score (AGHDA score>11) will also be re-tested following 6-months of growth hormone replacement therapy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Growth Hormone Deficiency (n=16): 16 asymptomatic GHD patients (who have confirmed GHD but who remain without GH replacement) will be compared with 16 healthy controls. Participants will be asked to undertake a single fasting blood sample and an MRI scan (whole body MRI and proton- and phosphorus-MR spectroscopy) to determine VAT, SAT and liver fat and muscle mitochondrial function. FGF21, body composition and mitochondrial function will be assessed in each of cohort to determine the correlation of FGF21 levels with VAT, SAT and liver fat.
- Healthy Controls (n=16): 16 healthy controls will be compared with 16 asymptomatic GHD patients (who have confirmed GHD but who remain without GH replacement). Participants will be asked to undertake a single fasting blood sample and an MRI scan (whole body MRI and proton- and phosphorus-MR spectroscopy) to determine VAT, SAT and liver fat and muscle mitochondrial function. FGF21, body composition and mitochondrial function will be measured in all cohorts to determine the correlation of FGF21 levels with VAT, SAT and liver fat.
- Growth Hormone Replacement Therapy (n=16): GHD patients, who are eligible for GH replacement therapy as part of their routine clinical care, according to the National Institute for Clinical Excellence (NICE) recommendations, based on the biochemical deficiency and the appropriate AGHDA questionnaire score (AGHDA score>11) will be recruited. These patients attend the Joint Endocrine clinic at University Hospital Aintree, Liverpool, and those who are about to commence growth hormone replacement will be asked to participate in this observational study.
  Anthropometric, biochemical including measurement of FGF21 and MR evaluation will be carried out in patients who are to be treated with GH as part of their routine clinical care immediately prior to GH therapy and after six months of replacement treatment. The type of GH and dose of treatment will be at the discretion of the treating physician. Standard doses will be used and patients will remain under the care of the supervising
  Interventions: Drug: Growth Hormone Replacement Therapy

INTERVENTIONS:
Drug: Growth Hormone Replacement Therapy — An observational study of patients who are commencing GH replacement as part of their routine NHS clinical care to assess changes in serum FGF21 concentration and determine how these relate to changes in body composition.
  Groups: Growth Hormone Replacement Therapy (n=16)

SUMMARY:
This study will recruit healthy controls (who have normal GH production and growth hormone levels) and patients identified as having GHD, who are deemed eligible for GH replacement therapy according to NICE guidelines. The patients recruited will have been identified as starting on GH by their referring clinicians and a decision made on their replacement therapy prior to their potential enrollment in the study. The study, or its research team, will have no influence on the decision as to whether a patient will start on GH, or on which of the many GH formulations that the patients receives. The proposed study is an observational study to determine how GH affects the plasma levels of Fibroblast growth factor 21 (FGF21) in response to treatment; and whether the change in FGF21 mirrors the improvement in body composition/fat deposition. FGF21 is a metabolic regulator that acts on multiple tissues to coordinate carbohydrate and lipid metabolism and regulate energy balance.

We hypothesize that FGF-21 is expressed and secreted from liver and skeletal muscle in humans in response to growth hormone administration and that levels may be reduced in patients with GHD compared with healthy controls. Furthermore, we believe that the beneficial effects of long-term GH replacement on body composition (reduction in visceral adipose tissue, subcutaneous adipose tissue and liver fat), on improvement in lipid profiles and on skeletal muscle mitochondrial function involve GH-induced release of FGF21.

DETAILED DESCRIPTION:
Growth hormone (GH) is involved in controlling people's general health and an underproduction of growth hormone (growth hormone deficiency or GHD) leads to people feeling generally unwell and having a lower feeling of well-being and quality of life scores. In addition, the investigators, and others, have demonstrated people with GHD have reduced muscle and bone strength and a greater storage of fat, particularly in unfavourable sites such as in the liver and within the abdomen (visceral fat), rather than beneath the skin (subcutaneous fat).

Treatment of GHD is achieved by administration of GH replacement therapy, given as a once daily subcutaneous injection, which generally reverses these symptoms. Due to its high cost, patients are only started on GH replacement depending on the impact that the GHD is having on their quality of life. Patients must be severely affected to be eligible for replacement therapy. Patients are screened for quality of life using a well validated, disease specific questionnaire (AGHDA, Adult Growth hormone deficiency questionnaire) and there are specific criteria that govern whether a patient with GHD warrants GH replacement and also whether they continue treatment (NICE guideline: Growth hormone deficiency (adults) - human growth hormone (TA64)).

This study will specifically determine whether the mechanism of action by which GH exerts its beneficial effects on metabolism (within adipose tissue and skeletal muscle) involves changes in serum FGF21 concentrations.

ELIGIBILITY:
All evaluations to determine eligibility into the study and for growth hormone replacement are performed as part of routine clinical care. It should be emphasised that no research specific screening tests will be performed. Patients deemed eligible for entry into study, who decline to participate in the research, will still be commenced on growth hormone in line routine clinical care.

Inclusion criteria: Patients with confirmed GH deficiency who are deemed eligible for GH replacement as assessed by the AGHDA QOL questionnaire.

Exclusion criteria: Claustrophobia or having significant metal work is a contra-indication to MRI scanning.

Withdrawal criteria: Patients will be withdrawn from the study if they discontinue their growth hormone replacement therapy for any clinical reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Secondary care clinic University advertisement
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Estimated); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
FGF21 | 6-months
  The primary outcome measure involves differences in serum FGF21 concentration between healthy controls and GHD patients, and changes in FGF21 concentration with GH replacement in patients with GHD

SECONDARY OUTCOMES:
Visceral and subcutaneous fat | 6-months
  Differences in visceral and subcutaneous fat volume between healthy controls and GHD patients.
  Changes in visceral and subcutaneous fat volume after 6 months of GH.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cuthbertson, PhD, Principal Investigator — University of Liverpool
Locations (2):
- United Kingdom (2):
  - MARIARC, Liverpool, Merseyside
  - University Hospital Aintree, Liverpool, Merseyside